CLINICAL TRIAL: NCT00373334
Title: A Double-Blind, Randomized, Parallel, Multicenter Study of Axid (Nizatidine) Oral Solution in the Treatment of Gastroesophageal Reflux Disease (GERD) Symptoms in Infants Age 30 Days-1 Year
Brief Title: Safety and Efficacy Study of Axid Use in Infants Suffering From Gastroesophageal Reflux Disease (GERD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Braintree Laboratories (Industry)
Responsible Party: John McGowan, Clinical Operations Manager, Braintree Laboratories, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BLI-AX-001
Record Dates: First submitted 2006-09-07; First posted 2006-09-08 (Estimated); Results first posted 2009-11-17 (Estimated); Last update posted 2009-11-18 (Estimated); Status verified 2009-11

CONDITIONS: Gastroesophageal Reflux Disease; GERD; Heartburn
Keywords: gastroesophageal reflux disease; GERD; heartburn
MeSH Terms: conditions — Gastroesophageal Reflux; Heartburn | interventions — Nizatidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: nizatidine (axid)
- 2 (Experimental)
  Interventions: Drug: nizatidine (axid)
- 3 (Sham Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: nizatidine (axid) — nizatidine (axid)
  Arms: 1
Drug: nizatidine (axid) — nizatidine (axid)
  Arms: 2
Drug: placebo — placebo
  Arms: 3

SUMMARY:
The objective of this study is to evaluate the efficacy, acceptability, and safety of Axid Oral Solution versus placebo in the treatment of gastroesophageal reflux disease (GERD) in infants age 30 days up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients age 30 days up to 1 year at Visit 1.
* Subjects must have a documented medical diagnosis of gastroesophageal reflux disease (GERD), confirmed by either endoscopy or pH monitoring, or by evaluation of baseline symptoms.
* Subjects must be greater than the 3rd percentile of weight and height for their age.
* Parents/guardians are competent and willing to provide consent and sign and date the institutional review board (IRB) approved consent form.
* Parents/guardians are willing to adhere to study requirements, including applying the conservative GERD management methods.
* Conservative GERD management methods have failed to adequately control GERD symptoms by Visit 2.
* Parent/guardian and infant live in the same household.
* Qualifying caregiver questionnaire score at Visits 1 & 2.

Exclusion Criteria:

* Any known esophageal disease or disorder, other than reflux esophagitis.
* Any active gastroduodenal ulceration, or clinical or endoscopic evidence of active gastrointestinal bleeding.
* Any prior esophageal or gastric surgery.
* Concurrent serious systemic disorders, including chronic respiratory disease, chronic neurologic disease, chronic renal disease, chronic liver disease.
* Subjects with clinically significant abnormal laboratory findings at screening.
* Premature infants < 37 weeks gestation at birth.
* Infants with prior neonatal intensive care unit admission for any reason.
* Hematemesis or apparent life-threatening events (ALTE).
* Concurrent treatment with any chronic medication except by permission of the study sponsor.
* Treatment with a histamine 2 receptor antagonist (H2RA), antacid, sucralfate, prostaglandin, or motility agent within 3 days before Visit 1; treatment with a proton pump inhibitor within 7 days before Visit 1.
* Requirement or likely requirement for a medical procedure or surgery during the study.
* Known hypersensitivity to an H2RA including nizatidine.
* Receipt of any investigational agent within the previous 30 days before randomization.
* Poor medical or psychiatric risks for therapy with an investigational drug, in the opinion of the investigator.
* Any condition in parent/guardian associated with poor subject compliance e.g., substance abuse); inability of parent/guardian to return for scheduled visits with their child.

Ages: 30 Days to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 138 (Actual)
Dates: Start 2006-08; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John McGowan, Study Director — Braintree Laboratories, Inc.
Locations (25):
- United States (25):
  - Hot Springs, Arkansas
  - Jonesboro, Arkansas
  - Little Rock, Arkansas
  - Searcy, Arkansas
  - Madiera, California
  - Centennial, Colorado
  - Orlando, Florida
  - Panama City, Florida
  - Tampa, Florida
  - Tifton, Georgia
  - Owensboro, Kentucky
  - Shreveport, Louisiana
  - Lincoln, Nebraska
  - Bismarck, North Dakota
  - Fargo, North Dakota
  - Fairfield, Ohio
  - Mason, Ohio
  - Hershey, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Clarksville, Tennessee
  - Houston, Texas
  - Missouri City, Texas
  - Temple, Texas
  - Ogden, Utah
  - South Jordan, Utah

RESULTS

PARTICIPANT FLOW:
Groups:
- Nizatidine 2.5 mg/kg Twice Daily: low dose nizatidine plus Conservative Measures
- Nizatidine 5.0 mg/kg Twice Daily: high dose nizatidine plus Conservative Measures
- Placebo: Placebo plus Conservative Measures
  Conservative Measures included:
  Hypoallergenic formula thickened with dry rice cereal Avoidance of seated and supine positioning Elimination of tobacco smoke exposure
Period: Overall Study
Arm/Group | Nizatidine 2.5 mg/kg Twice Daily | Nizatidine 5.0 mg/kg Twice Daily | Placebo
Started | 43 | 50 | 45
Completed | 33 | 32 | 32
Not Completed | 10 | 18 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nizatidine 2.5 mg/kg b.i.d. | Nizatidine 5.0 mg/kg b.i.d. | Conservative Measures Only | Total
Number analyzed (Participants) | 43 | 50 | 45 | 138
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 43 | 50 | 45 | 138
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 44 | 38 | 120
  Male | 5 | 6 | 7 | 18
Region of Enrollment [Number; unit: participants]
  United States | 43 | 50 | 45 | 138

OUTCOME MEASURES:

1. Primary Outcome: Infant Gastroesophageal Reflux Questionnaire Revised (I-GERQ-R) Success
Description: The I-GERQ-R contains 12 questions assessing gastroesophageal reflux disease (GERD) frequency and severity. A low I-GERQ-R score (minimum = 0) indicates minimal symptoms and a high I-GERQ-R score (maximum = 42) indicates more frequent and/or severe symptoms. Success is defined as a reduction in I-GERQ-R score of at least 5 points from baseline, provided a subject did not discontinue due to lack of efficacy or adverse event, and had been treated for at least 4 weeks.
Time Frame: 8 weeks
Population: The analysis population includes all patients that took drug and had any efficacy data reported. 5 patients that were lost to follow up (1 nizatidine 2.5 group, 1 nizatidine 5.0 group, 3 placebo group) were not included because they had no efficacy data and had not reported any adverse events.
Measure: Number; unit: participants
Arm/Group | Nizatidine 2.5 mg/kg b.i.d. | Nizatidine 5.0 mg/kg b.i.d. | Conservative Measures Only
Number analyzed (Participants) | 42 | 49 | 42
participants | 27 | 32 | 31
Statistical Analysis 1: Comparison: Nizatidine 5.0 mg/kg b.i.d. vs Conservative Measures Only; Test type: Superiority or Other; p = 0.528, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Nizatidine 2.5 mg/kg b.i.d. vs Conservative Measures Only; Test type: Superiority or Other; p = 0.341, Cochran-Mantel-Haenszel

2. Secondary Outcome: Investigator Assessment of Gastroesophageal Reflux Disease (GERD) Relief
Description: Subjective investigator assessment of GERD relief - rating categories were BETTER, NO CHANGE, or WORSE from baseline.
Time Frame: 8 weeks
Population: The analysis population includes all patients that took drug and reached the 8 week study timepoint.
Measure: Number; unit: participants
Arm/Group | Nizatidine 2.5 mg/kg b.i.d. | Nizatidine 5.0 mg/kg b.i.d. | Conservative Measures Only
Number analyzed (Participants) | 41 | 44 | 39
participants
  Better | 32 | 36 | 29
  No Change | 4 | 2 | 6
  Worse | 5 | 6 | 4
Statistical Analysis 1: Comparison: Nizatidine 2.5 mg/kg b.i.d. vs Conservative Measures Only; Comparison of nizatidine 2.5 group to placebo group. P-value is for overall difference between groups (not comparison of individual categories); Test type: Superiority or Other; p = 0.746, Chi-squared
Statistical Analysis 2: Comparison: Nizatidine 5.0 mg/kg b.i.d. vs Conservative Measures Only; Comparison of nizatidine 5.0 group to placebo group. P-value is for overall difference between groups (not comparison of individual categories); Test type: Superiority or Other; p = 0.262, Chi-squared

3. Secondary Outcome: Investigator Assessment of Gastroesophageal Reflux Disease (GERD) Severity
Description: Subjective investigator assessment of GERD severity - rating categories were NONE, MILD, MODERATE, or SEVERE.
Time Frame: 8 weeks
Population: The analysis population includes all patients that took drug and reached the 8 week study timepoint.
Measure: Number; unit: participants
Arm/Group | Nizatidine 2.5 mg/kg b.i.d. | Nizatidine 5.0 mg/kg b.i.d. | Conservative Measures Only
Number analyzed (Participants) | 41 | 44 | 38
participants
  None | 3 | 7 | 5
  Mild | 25 | 26 | 25
  Moderate | 10 | 9 | 7
  Severe | 3 | 2 | 1
Statistical Analysis 1: Comparison: Nizatidine 2.5 mg/kg b.i.d. vs Conservative Measures Only; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.609, Chi-squared
Statistical Analysis 2: Comparison: Nizatidine 5.0 mg/kg b.i.d. vs Conservative Measures Only; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.938, Chi-squared

ADVERSE EVENTS:
Arm/Group | Nizatidine 2.5 mg/kg b.i.d. | Nizatidine 5.0 mg/kg b.i.d. | Conservative Measures Only
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/50 | 1/45
Other Adverse Events (participants affected / at risk) | 27/43 | 31/50 | 31/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nizatidine 2.5 mg/kg b.i.d. (N=43) | Nizatidine 5.0 mg/kg b.i.d. (N=50) | Conservative Measures Only (N=45)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nizatidine 2.5 mg/kg b.i.d. (N=43) | Nizatidine 5.0 mg/kg b.i.d. (N=50) | Conservative Measures Only (N=45)
Diarrhea (Gastrointestinal disorders) | 4 | 4 | 5
Pyrexia (General disorders) | 6 | 1 | 3
Teething (Gastrointestinal disorders) | 4 | 3 | 3
bronchiolitis (Infections and infestations) | 3 | 6 | 2
conjunctivitis (Eye disorders) | 0 | 3 | 0
gastroenteritis (Infections and infestations) | 0 | 3 | 2
gastroesophageal reflux disease (Gastrointestinal disorders) | 2 | 10 | 4
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 4
otitis media (Infections and infestations) | 8 | 13 | 7
upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 13 | 6 | 15
vomiting (Gastrointestinal disorders) | 2 | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the principal investigator is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 360 days from the time submitted to the sponsor for review. The sponsor cannot extend the embargo.